CLINICAL TRIAL: NCT06083129
Title: Phase III Study Comparing GVHD Prophylaxis With ATG-thymoglobulin to ATLG-grafalon in Elderly Patients With Acute Myeloid Leukemia or Myelodysplasic Syndrome and Receiving an Allogeneic Hematopoietic Stem Cell Transplantation With a 10/10 HLA Matched Unrelated Donor Following a Reduced Intensity Conditioning Regimen by Fludarabine-treosulfan
Brief Title: Phase III Study Comparing GVHD Prophylaxis With ATG-thymoglobulin to ATLG-grafalon in Elderly Patients With Acute Myeloid Leukemia or Myelodysplasic Syndrome and Receiving an Allogeneic Hematopoietic Stem Cell Transplantation With a 10/10 HLA Matched Unrelated Donor
Acronym: OPTISAGE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: APHP230276
Record Dates: First submitted 2023-10-09; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-07

CONDITIONS: GVHD
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-T lymphocyte globulin (ATLG) (Active Comparator)
  Interventions: Drug: Grafalon
- Anti Thymocyte Globulins (ATG) (Active Comparator)
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Grafalon — 10 mg/Kg/day IV for 3 consecutive days (day-3 to -1 before transplantation)
  Arms: Anti-T lymphocyte globulin (ATLG)
Drug: Thymoglobulin — 2.5 mg/Kg/day IV for 2 consecutive days (day-3 and -2 before transplantation)
  Arms: Anti Thymocyte Globulins (ATG)

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) remains the only curative therapy in acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS). Most of the patients requiring an allo-HSCT are above 50 years of age and are transplanted with a reduced intensity conditioning (RIC) regimen. The optimal RIC and Graft Versus Host Disease (GVHD) prophylaxis regimen allowing a good control of the disease while preventing GVHD remains to be determined for elderly patients. A phase III trial comparing the conventional RIC fludarabine-busulfan 2 days to fludarabine-treosulfan demonstrated an advantage for the flu-treosulfan arm in terms of event free survival (EFS), that should therefore be considered as the new standard of RIC regimen for AML and MDS. GVHD prevention has a crucial role in post-transplant outcomes by potentially interfering with the graft-versus-leukemia (GVL) effect and immune reconstitution. Anti-thymocyte globulins (ATG) are recommended to reduce the risk of acute and chronic GVHD in transplants performed with matched unrelated donors. However, the optimal type of ATG between the 2 approved brands (ATG-thymoglobulin and ATLG-grafalon) displaying distinct characteristics and the optimal dose of ATG are still unknown. In a retrospective study of patients transplanted mainly with RIC with matched related and unrelated donors for haematological malignancies, we observed that Anti-T lymphocyte globulin (ATLG) was associated with a reduction of grade II-IV acute GVHD in comparison to ATG without increasing the incidence of relapse.

In this phase III randomised study, we propose to compare GVHD prevention with ATG versus ATLG in AML and MDS patients above 50 years of age transplanted with a matched unrelated donor following a fludarabine-treosulfan RIC, with the hypothesis that ATLG would better control GVHD in this population of patients thus limiting the risk of morbidity and mortality of the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 50 and ≤ 70 years
2. Patient between 50 and 55 years should be unfit for a myeloblative conditioning (SORROR score ≥2)
3. AML requiring allogeneic stem cell transplantation (intermediate or high-risk AML) in complete cytologic response (CR1 or above) or MDS requiring allogeneic stem cell transplantation (IPSS≥ 1.5 or IPSS-R > 4.5 or IPSS-R > 3-4.5 with risk features [rapide blast increase, life-threatening neutropenia (<0.3 G/L) or thrombopenia (<30G/L) or high transfusion needs (>2/month for 6 months)]
4. Without an HLA matched related donor
5. Having an identified matched HLA 10/10 unrelated donor
6. With usual criteria for HSCT:

   1. ECOG performans status ≤ 2
   2. No severe and uncontrolled infection
   3. Cardiac left ventricular ejection fraction ≥50%
   4. Lung DLCO > 40%
   5. Adequate organ function: ASAT and ALAT ≤ 3N, total bilirubin ≤ 2N, creatinine clearance ≥ 50 mL/min (except if those abnormalities are linked to the hematological disease)
7. With health insurance coverage
8. Having signed a written informed consent
9. Contraception methods must be prescribed during all the duration of the research

NB: The authorized contraceptive methods are:

* For women of childbearing age and in absence of permanent sterilization: oral, intravaginal or transdermal combined hormonal contraception, oral, injectable or transdermal progestogen-only hormonal contraception, intrauterine hormonal releasing system (IUS), sexual abstinence (only if this the preferred and usual lifestyle of the participants).
* For man in absence of permanent sterilization: sexual abstinence, condoms

Exclusion Criteria:

1. Cancer in the last 5 years (except basal cell carcinoma of the skin or "in situ" carcinoma of the cervix)
2. Uncontrolled infection
3. Seropositivity for HIV or HTLV-1 or active hepatitis B or C
4. Yellow fever vaccine and all others live virus vaccines within 2 months before transplantation
5. Heart failure according to NYHA (II or more) or Left ventricular ejection fraction < 50%.
6. Lung DLCO ≤ 40%
7. Preexisting acute hemorrhagic cystitis
8. Renal failure with creatinine clearance < 50ml / min
9. Pregnancy (β-HCG positive) or breast-feeding
10. Patients with any debilitating medical or psychiatric illness, which would preclude the realization of the SCT or the understanding of the protocol
11. Patient under state medical aid
12. Patient under legal protection (protection of the court, or in curatorship or guardianship).
13. For Grafalon: Hypersensitivity to the active substance or to any of the excipients
14. For Thymoglobulin: Hypersensitivity to rabbit proteins or to any of the excipients
15. Participation in other interventional clinical trials
16. Any contraindication mentioned in the SmPC of all auxiliary medicinal products planned to be used in the trial: cyclosporine, mycophenolate mofetil, fludarabine, treosulfan

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade II-IV acute Graft Versus Host Disease (GVHD) according to the Mount Sinai Acute GVHD International Consortium (MAGIC) classification | At day 100 post-transplantation
  Acute GVHD MAGIC classification permit to diagnose and score the severity of acute GVHD.
  MAGIC score varies from Grade 0 to Grade 4. The higher the score the more severe the damage.

SECONDARY OUTCOMES:
Number of patients with at least 3 consecutive days with neutrophils > 0.5 G/L and platelets > 20 G/L | Up to 24 months
  Hematopoietic recoveries
T, B, NK, regulatory T cell and gammaglobulin levels in the peripheral blood | 1 month after transplantation
  Immune reconstitution
T, B, NK, regulatory T cell and gammaglobulin levels in the peripheral blood | 100 days after transplantation
  Immune reconstitution
T, B, NK, regulatory T cell and gammaglobulin levels in the peripheral blood | 6 months after transplantation
  Immune reconstitution
T, B, NK, regulatory T cell and gammaglobulin levels in the peripheral blood | 12 months after transplantation
  Immune reconstitution
T, B, NK, regulatory T cell and gammaglobulin levels in the peripheral blood | 24 months after transplantation
  Immune reconstitution
Percentage of chimerism | 1 month after transplantation
Percentage of chimerism | 100 days after transplantation
Percentage of chimerism | 6 months after transplantation
Percentage of chimerism | 12 months after transplantation
Incidence of grade I acute GVHD | Up to 24 months
  Treatments for acute GVHD will be described : first line treatment, response to steroids, treatment courses for refractory acute GVHD
Incidence of chronic GVHD | 12 months after transplantation
  Incidence of chronic GVHD according to National Institutes of Health (NIH) classification. The gradation of chronic GvHD is defined by the number and score of affected organ. The higher the score of each organ and the higher the number of organs affected, the more severe the damage.
Incidence of chronic GVHD | 24 months after transplantation
  Incidence of chronic GVHD according to National Institutes of Health (NIH) classification. The gradation of chronic GvHD is defined by the number and score of affected organ. The higher the score of each organ and the higher the number of organs affected, the more severe the damage.
Incidence of relapse | 12 months after transplantation
  Relapse will be defined by the reappearance of leukemic cells or MDS features after allo-HSCT in the bonne marrow (cytology +/- cytogenetic analysis from bone marrow aspiration) or extra-medullary sites (proven by a biopsy).
Incidence of relapse | 24 months after transplantation
  Relapse will be defined by the reappearance of leukemic cells or MDS features after allo-HSCT in the bonne marrow (cytology +/- cytogenetic analysis from bone marrow aspiration) or extra-medullary sites (proven by a biopsy).
Progression free survival | 12 months after transplantation
Progression free survival | 24 months after transplantation
Number of severe infections | 100 days after transplantation
  Severe infections correspond to grade 3-4 according to Common Terminology Criteria for Adverse Events
Number of severe infections | 12 months after transplantation
  Severe infections correspond to grade 3-4 according to Common Terminology Criteria for Adverse Events
Incidence of CytoMegaloVirus (CMV) reactivation | 100 days after transplantation
Incidence of CytoMegaloVirus (CMV) reactivation | 6 months after transplantation
Incidence of CytoMegaloVirus (CMV) reactivation | 12 months after transplantation
Incidence of Ebstein Barr Virus (EBV) reactivation | 100 days after transplantation
Incidence of Ebstein Barr Virus (EBV) reactivation | 6 months after transplantation
Incidence of Ebstein Barr Virus (EBV) reactivation | 12 months after transplantation
Non-relapse mortality | 6 months after transplantation
Non-relapse mortality | 12 months after transplantation
Non-relapse mortality | 24 months after transplantation
Overall survival | 12 months after transplantation
Overall survival | 24 months after transplantation
GVHD and relapse free survival (GRFS) | Up to 24 months after transplantation
  Defined by being alive without disease relapse and without having developed acute grade III-IV or severe chronic GVHD
Health-related Quality of life | At inclusion
  Assessed by using the FACT-BMT-v4 questionnaire. It is a 50 items score. The score varies between 0 to 200. The higher the score the lower the quality of life.
Health-related Quality of life | 100 days after transplantation
  Assessed by using the FACT-BMT-v4 questionnaire. It is a 50 items score. The score varies between 0 to 200. The higher the score the lower the quality of life.
Health-related Quality of life | 6 months after transplantation
  Assessed by using the FACT-BMT-v4 questionnaire. It is a 50 items score. The score varies between 0 to 200. The higher the score the lower the quality of life.
Health-related Quality of life | 12 months after transplantation
  Assessed by using the FACT-BMT-v4 questionnaire. It is a 50 items score. The score varies between 0 to 200. The higher the score the lower the quality of life.
Number of days of hospitalization for the transplant and after the hospitalization for transplantation related complications | Up to 12 months after transplantation
Incidence and severity of veino-occlusive disease (VOD) | 100 days after transplantation
Lymphocyte counts on standard blood counts before conditioning | 7 days before transplantation
Number of late acute GvHD, overlap syndromes and chronic GvHD | from day 100 to day 120 after transplantation

IPD SHARING:
Plan to Share IPD: Undecided